CLINICAL TRIAL: NCT03555552
Title: Point of Care Testing to Improve Monitoring of LVAD Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00089633
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Anticoagulation and Thrombosis Point of Care Test (AT-POCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anticoagulation and Thrombosis Point of Care Test (AT-POCT) (Experimental)
  Interventions: Device: Anticoagulation and Thrombosis Point of Care Test(AT-POCT); Device: Duke Central Automated Laboratory (DCAL)
- Duke Central Automated Laboratory (DCAL) (Active Comparator)
  Interventions: Device: Anticoagulation and Thrombosis Point of Care Test(AT-POCT); Device: Duke Central Automated Laboratory (DCAL)

INTERVENTIONS:
Device: Anticoagulation and Thrombosis Point of Care Test(AT-POCT) — Capillary action automatically draws blood into the channel containing printed assay reagents which solubilize upon contact with blood and react with analytes of interest.
Device: Duke Central Automated Laboratory (DCAL) — DCAL measurement of INR will occur by an ACL TOP 750 Analyzer (IL Inc.), and LDH by standard enzymatic activity assay will be run on the automated Beckman DxC800.

SUMMARY:
The purpose of this study is to develop and validate the accuracy of a low-cost "point-of-care" test (POCT) that allows monitoring of markers for anticoagulation and thrombosis (local coagulation or clotting of the blood), to be used by patients with advanced heart failure (AHF) on left ventricular assist device (LVAD) support. The investigators central hypothesis is that the fully-printed AT-POCT utilizing low-cost (printed) cassettes and detector will produce an inexpensive and convenient option for daily self-monitoring of PT/INR and LDH over existing methods.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Subject has signed Informed Consent Form (ICF)
* For LVAD patient cohort, they are on LVAD support from 2 weeks to 10 years.

Exclusion Criteria:

* Patients with dementia, altered mental status, any psychiatric condition or mental disability that would prohibit the understanding or rendering of informed consent are not eligible
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Interclass correlation between PT/INR and LDH measurements | 1 study day
  The primary outcome is acceptable inter-rater agreement between our measure and the clinical gold standards for both PT/INR and LDH. This will be defined as an interclass correlation of > 0.8 with a CI lower bound of 0.1 based on the sample size of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Chilkoti, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No